CLINICAL TRIAL: NCT01673776
Title: Can a Multimodal Approach Improve the Outcome of Patients With a Proximal Femoral Fracture?
Brief Title: Multimodal Approach to Improve the Outcome of Patients With a Proximal Femoral Fracture
Acronym: FEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMO
Record Dates: First submitted 2012-08-20; First posted 2012-08-28 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Proximal Femoral Fracture
Keywords: Proximal femoral fracture; multimodal intervention; goal directed therapy (GDT); hemodynamic intervention; outcome
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- K group (No Intervention): commonly used therapy
- M group (Experimental): multimodal intervention
  Interventions: Device: PulsioFlex® Monitoring

INTERVENTIONS:
Device: PulsioFlex® Monitoring — * goal directed therapy according to PulsioFlex® Monitoring- measurements
  * femoral catheter
  * extended perioperative monitoring
  * nutritional supplementation, (if necessary)
  Arms: M group

SUMMARY:
This study is designed to compare the outcome of patients with proximal femoral fractures with different perioperative regimes: a group with a multimodal intervention and a control group.

DETAILED DESCRIPTION:
Femoral neck fractures constitute both a social and economic challenge. The one year mortality of affected patients amounts to 33%, wherein cardio-vascular complications are the major contributor. It is an objective of the present study to investigate whether a multi-modal perioperative intervention can improve the outcome of these patients.

We plan to carry out a prospective randomized controlled clinical study. Patients with an age above 60 years and proximal femoral fractures (femoral neck fractures or pertrochanteric femoral fractures) are to be included. These are divided into two groups, K and M. General anaesthesia is applied to both groups. In group K a commonly used therapy will be applied whereas in group M an intesified perioperative care will be carried out. The objectives are to provide sufficient analgesia, normotonia and normothermia. Hence, a femoral catheter is applied for pain therapy already preoperatively. Moreover, the pulmonal situation is improved by means of oxygen as needed. The cardiovascular situation is evaluated and optimized by means of extended hemodynamic monitoring both pre- and postoperatively. If needed, the nutrition of the patients is supplemented with highly caloric drinks.

A primary common endpoint is the appearance of postoperative complications. These include cardiovascular, cerebrovascular, pulmonal, renal and surgical complications. Secondary endpoints are mortality, duration of the stay at the hospital and intensive care duration. It is the objective of the study to reduce the probability for at least one postoperative complication from 50% to 25% (α=0,05 and 1-β=0,80). To this end 132 patients would have to be included in the study.

All participants are to be contacted by phone one year after the surgery and their health situation is to be determined.

ELIGIBILITY:
Inclusion Criteria:

* proximal femoral fracture (femoral neck fracture/ pertrochanteric femoral fracture)
* Age ≥ 60 years
* written informed consent

Exclusion Criteria:

* pathological fracture
* multiple trauma
* fracture during a hospital stay due to a different disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
postoperative complications | The participants will be followed for the duration of hospital stay, an expected average of 14 days
  postoperative complications: cardiovascular, cerebrovascular, pulmonal, renal and surgical complications

SECONDARY OUTCOMES:
mortality | 1 year
duration of the stay at the hospital | 1 year
intensive care duration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Pedersen SJ, Borgbjerg FM, Schousboe B, Pedersen BD, Jorgensen HL, Duus BR, Lauritzen JB; Hip Fracture Group of Bispebjerg Hospital. A comprehensive hip fracture program reduces complication rates and mortality. J Am Geriatr Soc. 2008 Oct;56(10):1831-8. doi: 10.1111/j.1532-5415.2008.01945.x. PMID 19054201
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Derived] Schmid S, Blobner M, Haas B, Lucke M, Neumaier M, Anetsberger A, Jungwirth B. Perioperative multi-system optimization protocol in elderly hip fracture patients: a randomized-controlled trial. Can J Anaesth. 2019 Dec;66(12):1472-1482. doi: 10.1007/s12630-019-01475-9. Epub 2019 Sep 17. PMID 31531828